CLINICAL TRIAL: NCT03922035
Title: A Randomized Open Label Pilot Study of Clostridium Butyricum MIYAIRI 588 (CBM588) in Recipients of Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: CBM588 in Improving Clinical Outcomes in Patients Who Have Undergone Donor Hematopoietic Stem Cell Transplant
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18193; NCI-2018-01886 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18193 (Other: City of Hope Medical Center)
Record Dates: First submitted 2018-09-10; First posted 2019-04-19 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (CBM588) (Experimental): Patients receive standard peri-/post-transplant supportive care and CBM588 PO BID from day of admission to day 28 in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Best Practice; Drug: Clostridium butyricum CBM 588 Probiotic Strain
- Arm II (standard of care) (Active Comparator): Patients receive standard peri-/post-transplant supportive care.
  Interventions: Other: Best Practice

INTERVENTIONS:
Other: Best Practice — Receive standard peri-/post-transplant supportive care
  Other Names: standard of care; standard therapy
Drug: Clostridium butyricum CBM 588 Probiotic Strain — Given PO
  Other Names: C. butyricum CBM 588 Probiotic Strain; C. butyricum MIYAIRI Strain; C. butyricum Strain MIYAIRI 588; CBM 588; CBM588; Clostridium butyricum MIYAIRI 588; Clostridium butyricum MIYAIRI 588 Probiotic Strain; MIYAIRI 588; MIYAIRI 588 Strain of C. butyricum
  Arms: Arm I (CBM588)

SUMMARY:
This pilot trial studies the side effects and how well CBM588 works in improving clinical outcomes in patients who have undergone donor hematopoietic stem cell transplant. Gut microbiota (formerly called gut flora) is the name given to the microbe (bacteria) population living in the intestine. Gut bacteria help the body to digest certain foods that the stomach and small intestine have not been able to digest. CBM588, may increase gut bacteria biodiversity, prevent recurrent symptoms of gastrointestinal toxicity (ranging from diarrhea to life-threatening inflammation of the colon).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. In patients with hematologic malignancies who are undergoing standard reduced intensity conditioning regimen (RIC) prior to allogeneic stem cell transplantation, to evaluate the safety and feasibility of Clostridium butyricum CBM 588 probiotic strain (CBM588) treatment by assessing:

Ia. Type, frequency, severity, attribution, time course and duration of adverse events, including diarrhea, bloodstream/intestinal infections.

Ib. Patient compliance, the patients' ability to take CBM588 during the treatment period.

SECONDARY OBJECTIVES:

I. Compare the incidence and severity of adverse events (AE) among CBM588-treated and untreated patients, including diarrhea, bloodstream infections and intestinal infections.

II. Estimate overall survival (OS), cumulative incidence (CI) of chronic graft versus host disease (GVHD), relapse/progression, and non-relapse mortality (NRM) at 100 days, 6 months, 1 year and 2 years.

EXPLORATORY OBJECTIVES:

I. Compare gut microbiome diversity among CBM588-treated/untreated patients. II. Obtain a preliminary estimate of the possible association between gut microbiome diversity and bloodstream infections.

III. Characterize and compare graft versus host disease (GVHD) inflammatory biomarkers (presence, level) among CBM588-treated and untreated patients.

IV. Obtain preliminary estimates of gut microbiome diversity, as assessed by the inverse Simpson Index, in CBM588-treated/untreated patients.

V. Obtain a preliminary estimate of the possible association between gut microbiome diversity and acute GVHD cumulative incidence, including time to onset.

VI. Characterize and compare urinary uindoxyl sulfate, tryptophan and kynurenine levels between CBM588- treated and untreated patients.

VII. To obtain a preliminary estimate of gut microbiome diversity and calorie intake.

VIII. Characterize and compare impact of CBM588 administration on regulatory T cells (T regs) reconstitution between CBM588-treated and untreated patients.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (CBM588): Patients receive standard peri-/post-transplant supportive care and CBM588 orally (PO) twice daily (BID) from day of admission to day 28 in the absence of disease progression or unacceptable toxicity.

ARM II (STANDARD OF CARE): Patients receive standard peri-/post-transplant supportive care.

After completion of study treatment, patients are followed up for 100 days and then up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative.

  * Assent, when appropriate, will be obtained per institutional guidelines.
* Willingness to be followed for the planned duration of the trial (2 years).
* Karnofsky performance status must be >= 60%.
* Any hematologic disorders receiving allogeneic hematopoietic stem cell transplant with reduced intensity conditioning.
* Planned 8/8 or 7/8 (human leukocyte antigens [HLA]-A, B, C, DR) related or unrelated donor hematopoietic cell transplantation (HCT).
* Clinical Laboratory and Organ Function Criteria: Consistent with City of Hope (COH) standard operating procedure (SOP) for "patient evaluation for selection for hematopoietic cell transplantation.
* Patient is eligible to receive allogeneic hematopoietic cell transplantation with reduced intensity conditioning.
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 3 months after the last dose of protocol therapy.

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only).

Exclusion Criteria:

* Failure of research participant to understand the basic elements of the protocol and/or the risks/benefits of participating in this pilot study. A legal guardian may substitute for the research participant.
* Refusing to use contraception up to 90 days post-HCT.
* Pregnant and/or breast feeding if a female recipient.
* Patients with history of chronic intestinal disease (e.g., Crohn's disease, ulcerative colitis).
* In the opinion of the principal investigator (PI), the participant has a condition that will preclude them from complying with study treatment.
* Research participants receiving any other investigational agents.
* Known or documented history of hypersensitivity to all the listed antibiotics, used for severe infections related to CBM588:

  * Ampicillin.
  * Chloramphenicol.
  * Clindamycin.
  * Erythromycin.
  * Metronidazole.
  * Tetracycline.
  * Vancomycin.
* Research participants with presence of other active malignancy within 2 years of study entry. Participants with history of prior malignancy treated with curative intent who achieved complete response (CR) more than 2 years before study entry are eligible. This exclusion rule does not apply to non-melanoma skin tumors and in-situ cervical cancer.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent (i.e., research participants whom are severe lactose intolerance or intolerance to milk products).
* Research participants having any uncontrolled illness including ongoing or active infection. Research participants with known active hepatitis B or C infection; research participants who are human immunodeficiency virus (HIV) seropositive based on testing performed within 4 weeks of enrollment; research participants with any signs or symptoms of active infection, positive blood cultures, or radiological evidence of infections.
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures.
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2026-03-04 (Estimated); Study Completion 2026-03-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | From initiation of treatment until end of treatment assessed up to 100 days
  Will be scored according to the modified Bearman Scale and National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5 scale. Observed toxicities will be summarized in terms of type (organ affected or laboratory determination), severity, time of onset, duration, probable association with the study treatment and reversibility or outcome.
Feasibility of CBM588 | During the safety lead-in phase
  Will be evaluated by assessment of patients' ability to take half of the specified dose.

SECONDARY OUTCOMES:
Incidence and severity of adverse events | Up to 2 years
  Assessed by modified Bearman criteria and NCI CTCAE version 5 scale. Will be compared among CBM588 treated and untreated patients.
Overall survival | Up to 2 years
  Will be estimated using the product-limit method of Kaplan and Meier.
Cumulative incidence (CI) of chronic graft versus host disease (cGVHD) | Up to 2 years
  Will be estimated using the method described by Gooley et al (1999).
CI of acute graft versus host disease (aGVHD) | Up to 2 years
  Will be estimated using the method described by Gooley et al (1999).
CI of relapse/progression of disease | Up to 2 years
  Will be estimated using the method described by Gooley et al (1999).
Non-relapse mortality | Up to 2 years
  Will be estimated using the method described by Gooley et al (1999).

OTHER OUTCOMES:
Gut microbiome diversity | Up to 2 years
  Will be assessed by the inverse Simpson index. Will be compared among CBM588-treated/untreated patients and assessed by Fisher's exact test or two-sample Wilcoxon test whenever appropriate.
Gut microbiome diversity and bloodstream infection | Up to 2 years
  Incidence of bloodstream infections and infectious enterocolitis will be evaluated and a preliminary estimate of the association between gut microbiome diversity and blood stream infections will be obtained.
Gut microbiome diversity aGVHD incidence | Up to 2 years
  Will be obtained based on: 1) evaluation and comparison of presence and levels GVHD/inflammatory biomarkers including TNFR1, ST2, Reg3 alpha, TNF-alpha, IL-8 and TGF-beta 1 between the 2 study arms, and 2) incidence, site (gastrointestinal [GI], liver, and skin), severity (grade III-IV GI toxicity per the NCI CTCAE version 5 Scale) and time to onset of aGVHD among treated and untreated patients.
Levels of tryptophan metabolites | Up to 2 years
  Presence and levels of urinary uindoxyl sulfate, tryptophan and kynurenine (markers of GI GVHD complications) will be evaluated and compared between CBM588-treated and untreated patients.
Impact on regulatory T cells (T regs) | Up to 2 years
  Presence and levels T regs will be evaluated and compared in blood samples from patients among treated and untreated patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ryotaro Nakamura, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States